CLINICAL TRIAL: NCT07379775
Title: Evaluation of the Reliability of Anterior Active Rhinomanometry as an Independent Tool for Surgical Indication in Nasal Obstruction
Brief Title: Evaluation of the Reliability of AAR as an Independent Tool for Surgical Indication in Nasal Obstruction
Acronym: RHINOVE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-CHITS-018
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with nasal obstruction: Patients scheduled for surgery who underwent preoperative rhinomanometry
  Interventions: Procedure: preoperative rhinomanometry

INTERVENTIONS:
Procedure: preoperative rhinomanometry — The performance of AAR requires a pressure sensor placed within a facial mask to measure the pressure at the entrance of the ventilated nasal cavity. Another sensor is placed in the nasal vestibule of the contralateral nasal cavity to extrapolate the pressure at the exit of the ventilated nasal cavity. Measurements are therefore performed alternately on the right and left sides, but never on both sides simultaneously.
  AAR can be performed at rest in the seated position after 20 min in the supine position, or during forced inspiration.
  In our practice, AAR is performed without the use of nasal decongestants.
  Normal values of nasal resistance measured by rhinomanometry are as follows:
  * Uninasal resistance ≤ 6 cmH₂O/L/s (or 0.6 Pa/cm³/s);
  * Binasal resistance ≤ 3 cmH₂O/L/s (or 0.3 Pa/cm³/s);
  * Uninasal resistance ≥ 0.6 Pa/cm³/s, with or without vasoconstrictor, suggests septal deviation;
  * Binasal resistance after VC ≥ 0.3 Pa/cm³/s suggests bilateral inferior turbinate hypertrophy

SUMMARY:
Nasal obstruction (NO) affects ~30% of the population and is a very common reason for consultation in otorhinolaryngology (ORL). In the majority of cases, the origin is inflammatory (allergic rhinitis and chronic rhinosinusitis) while in a minority of cases, the origin is structural, including septal deviation and inferior turbinate hypertrophy.

NO significantly impairs patients' quality of life (QoL) and olfactory performance and also represents a contributing factor and comorbidity in asthma and obstructive sleep apnea syndrome. Several questionnaires for assessing QoL are available and routinely used to evaluate the impact of NO on patients : VAS, NOSE score, SNOT-22, and RhinoQOL score.

Several objective functional methods for assessing NO have been described : acoustic rhinometry, nasal peak inspiratory flow, and active rhinomanometry. Rhinomanometry is a simple, non-invasive functional assessment method that allows for objective and quantitative analysis of nasal airway patency, thereby complementing the clinical and imaging evaluation of NO.

It has been recommended for the diagnosis of NO in cases of chronic rhinitis and chronic rhinosinusitis with nasal polyposis. Rhinomanometry comprises anterior active (AAR), posterior, and per-nasal rhinomanometry. AAR is the most commonly used method and is the only technique routinely available to clinicians. AAR provides precise information regarding the presence of nasal resistance responsible for NO. However, it should not be used as a standalone diagnostic tool due to its poor correlation with QoL questionnaires such as VAS and NOSE.

Whether used alone or in combination with nasal decongestants, AAR provides a high predictive value for the outcomes of septoplasty and laser-assisted turbinoplasty.

When surgery is indicated, its performance depends on:

* type of obstruction or anatomical abnormality identified on clinical examination and/or computed tomography and/or AAR;
* patient's symptoms and impairment of QoL NOSE and SNOT-22;
* failure of a well-conducted first-line medical nasal treatment. Thus, in cases of septal deviation, septoplasty is performed; in cases of inferior turbinate mucosal hypertrophy with failure of medical treatment, turbinoplasty is performed; and in cases of mixed lesions, septo-turbinoplasty is performed.

However, the concordance rate between the surgical technique indicated by clinical examination and computed tomography and the indications suggested by AAR is only 48.5%.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older with nasal obstruction (NO).
2. Patients scheduled for surgery: septoplasty ± turbinoplasty ± rhinoplasty for nasal obstruction.
3. Patients who have undergone a preoperative rhinomanometry assessment.
4. Patients consented to participation

Exclusion Criteria:

1. Nasal polyps.
2. Chronic edematous-purulent rhinosinusitis (e.g., cystic fibrosis).
3. Crusting rhinosinusitis (e.g., sarcoidosis, granulomatosis with polyangiitis [Wegener's]).
4. Current or previously treated nasal or sinus tumors, or patients undergoing tumor work-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with nasal obstruction, scheduled for surgery, and having undergone preoperative rhinomanometry
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the reliability of an abnormal (vs. normal) binary result of preoperative anterior active rhinomanometry as an independent tool for confirming the indication for endonasal surgery in patients presenting with nasal obstruction. | the day of surgery
  The result was considered normal if: Uninasal resistance ≤ 6 cmH₂O/L/s (or 0.6 Pa/cm³/s); Binasal resistance ≤ 3 cmH₂O/L/s (or 0.3 Pa/cm³/s). The criteria is 1) Percentage of patients with an abnormal versus normal preoperative AAR result; and 2) calculation of the positive and negative predictive values (PPV and NPV) of AAR as an independent tool for confirming surgical indication.

SECONDARY OUTCOMES:
To evaluate the correlation between the preoperative NOSE score and a preoperative AAR considered abnormal. | preoperative visit
  Correlation coefficient between the preoperative NOSE score and the preoperative AAR result (normal/abnormal).
To evaluate the correlation between the preoperative SNOT-22 score and a preoperative AAR considered abnormal. | preoperative visit
  Correlation coefficient between the preoperative SNOT-22 score and the preoperative AAR result (normal/abnormal)
To assess the improvement in patients' quality of life at 3 months postoperatively using the NOSE score in patients with a preoperative AAR considered abnormal | 3 months after surgery
  Difference between pre- and 3-month postoperative NOSE scores in patients with an abnormal preoperative AAR result
To assess the improvement in patients' quality of life at 3 months postoperatively using the SNOT-22 score in patients with a preoperative AAR considered abnormal | 3 months after surgery
  Difference between pre- and 3-month postoperative SNOT-22 scores in patients with an abnormal preoperative AAR result
To assess the improvement in AAR at 3 months postoperatively in patients with a preoperative AAR considered abnormal | 3 months after surgery
  Percentage of AAR results significantly improved at 3 months postoperatively in patients with an abnormal preoperative AAR
To assess the improvement in the apnea-hypopnea index (AHI) at 3 months postoperatively in patients with identified obstructive sleep apnea and a preoperative AAR considered abnormal | 3 months after surgery
  Difference between pre- and 3-month postoperative apnea-hypopnea index (AHI) in patients with identified sleep apnea and an abnormal preoperative AAR result
To assess the improvement in continuous positive airway pressure (CPAP) adherence at 3 months postoperatively in patients with identified obstructive sleep apnea and a preoperative AAR considered abnormal. | 3 months after surgery
  Difference between pre- and 3-month postoperative adherence to continuous positive airway pressure (CPAP) in patients with identified sleep apnea and an abnormal preoperative AAR result.

CONTACTS AND LOCATIONS:
Overall Officials: Heritsilavo Eloi RAMILISON, MD, Study Director — Centre Hospitalier de la Dracénie - Draguignan
Locations (1):
- Centre Hospitalier de la Dracénie, Draguignan, Var, France

IPD SHARING:
Plan to Share IPD: No